CLINICAL TRIAL: NCT04027400
Title: Effects of Computer-Assisted Cognitive Rehabilitation Programs With Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19959
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Cognitive Impairment; Breast Cancer
Keywords: survivor; cognitive rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: two groups with different treatment
Who Masked: Participant
Masking Description: Participants never told which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primarily visual computer exercises (Active Comparator): Participant performs visual computer exercises 30 minutes a day, five days a week for one month.
  Interventions: Behavioral: computer-assisted rehabilitation
- Visual+Audio (Experimental): Participant performs audio computer exercises and some visual computer exercises 30 minutes a day, five days a week for one month
  Interventions: Behavioral: computer-assisted rehabilitation

INTERVENTIONS:
Behavioral: computer-assisted rehabilitation — Participant is presented with 10 exercises a day, 3 minutes each. When participant achieves 100% accuracy of the exercise, he/she gets a higher level of exercise. Levels of range from 1-9. Exercises are changed every week by researcher.
  Other Names: visual and audio computer exercises

SUMMARY:
Potential study participants will be recruited at breast cancer survivor support groups. Informed consent will be obtained with a form approved by the TWU IRB and participants will complete 4 tests. Then participants will be randomly assigned to one of two computer-assisted cognitive programs. Participants will be sent by email, exercises specific to their assigned computer-assisted cognitive program from Happyneuron Pro (http://ie.scientificbraintrainingpro.eu/). Cognitive training on the computer entails 30 minutes a day, five times a week for one month. At the end of the study, the four pretests will be repeated, a satisfaction survey administered.

DETAILED DESCRIPTION:
Potential study participants will be recruited using a recruitment script and recruitment brochure at breast cancer survivor support groups. Participants recruited to the study will be contacted to set up a pre-test data collection session. Prior to any testing, informed consent will be obtained with a form approved by the TWU IRB. After informed consent is obtained participants will complete tests of Digit Span Task, FACT-Cognitive Function (Version 3), Quality of Life Patient/Cancer Survivor Version and Engagement in Meaningful Activities Survey, and issued a tablet if they prefer. Then participants will be randomly assigned to one of two computer-assisted cognitive programs. Participants will be sent by email, exercises specific to their assigned computer-assisted cognitive program from Happyneuron Pro (http://ie.scientificbraintrainingpro.eu/). Cognitive training on the computer entails 30 minutes a day, five times a week for one month. 6. At the end of the study, the four pretests will be repeated, a satisfaction survey administered, and any issued tablets collected. Pre and post testing, obtaining of written consent, and issuing and returning a tablet will occur at the support group location. If this location is not available, they will occur at TWU in a quiet room. If TWU is not convenient to the participant, a quiet location that is suitable to maintain confidentiality for the participant will be chosen in collaboration with the participant.

ELIGIBILITY:
Inclusion Criteria:

* study participant self-identifies as breast cancer survivor
* had treatment that may have included surgery, chemotherapy, radiation, pharmacological or any combination of these treatments
* participant states has cognitive problems due to cancer treatment

Exclusion Criteria:

* persons who cannot read or understand spoken English
* have disorders that may affect their cognition including major mental disorder, central nervous system disorders, Alzheimer's disease, dementia, developmental delay, traumatic brain injury, or cerebrovascular accident.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-02-25 (Estimated); Study Completion 2020-02-26 (Estimated)

PRIMARY OUTCOMES:
Digit span | 10 minutes
  Working memory was measured by the digit span, shown to discriminate between BCS and controls.19 It takes approximately 10 minutes to administer and has high reliability (.891) for forward span and low for backwards span (.598).
FACT-COG | 10 minutes
  The FACT-COG contains 4 subscales of perceived cognitive impairment, comments from others, perceived cognitive abilities, and impact of cognition on quality of life which are summed to provide a score. Fact-Cog demonstrates acceptable test-retest reliability (.707) and validity (.762)
CANCER PATIENT/CANCER SURVIVOR VERSION | 10 minutes
  Quality of life as it relates to cancer survival, was measured with the 41 item Quality of Life Instrument (CANCER PATIENT/CANCER SURVIVOR VERSION).21 The overall QOL-CS tool test re-test reliability is .89
EMAS | 10 minutes
  Frequency of engagement in meaningful activities was assessed with the Engagement in Meaningful Activities Survey (EMAS) to calculate how often a subject participates in 12 activities.

SECONDARY OUTCOMES:
Satisfaction Survey | 5 minutes
  3 questions delivered post intervention on participant satisfaction with being in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa M Smith, PhD, Principal Investigator — Associate Professor
Locations (1):
- Texas Woman's University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No